CLINICAL TRIAL: NCT00787605
Title: An 8-week Study to Evaluate the Efficacy and Safety of Aliskiren HCTZ (300/25 mg) Compared to Amlodipine (10 mg) in Patients With Stage 2 Systolic Hypertension and Diabetes Mellitus
Brief Title: Aliskiren HCTZ Compared to Amlodipine in Patients With Stage 2 Systolic Hypertension and Diabetes Mellitus
Acronym: ASTRIDE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: External Affairs, Novartis
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CSPP100A2409
Record Dates: First submitted 2008-11-05; First posted 2008-11-07 (Estimated); Results first posted 2011-05-23 (Estimated); Last update posted 2016-10-27 (Estimated); Status verified 2011-05

CONDITIONS: Hypertension; Diabetes Mellitus
Keywords: Hypertension, diabetes mellitus, aliskiren, hydrochlorothiazide, systolic blood pressure, diastolic blood pressure, amlodipine, stage 2
MeSH Terms: conditions — Hypertension; Diabetes Mellitus | interventions — Amlodipine; Hydrochlorothiazide; aliskiren

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Amlodipine (Active Comparator): Amlodipine 5 mg for 1 week followed by Amlodipine 10 mg for 7 weeks
  Interventions: Drug: Amlodipine
- Aliskiren / HCTZ (Experimental): Aliskiren / HCTZ 150/12.5 mg for 1 week followed by 300/25 mg for 7 weeks
  Interventions: Drug: Hydrochlorothiazide (HCTZ); Drug: Aliskiren

INTERVENTIONS:
Drug: Amlodipine — Amlodipine 5 mg for 1 week followed by Amlodipine 10 mg for 7 weeks
  Arms: Amlodipine
Drug: Hydrochlorothiazide (HCTZ) — Hydrochlorothiazide 12.5 mg for 1 week followed by Hydrochlorothiazide 25 mg for 7 weeks
  Arms: Aliskiren / HCTZ
Drug: Aliskiren — Aliskiren 150 mg for 1 week followed by Aliskiren 300 mg for 7 weeks
  Arms: Aliskiren / HCTZ

SUMMARY:
The purpose of the study is to evaluate the blood pressure lowering effect and safety of aliskiren in combination with Hydrochlorothiazide (HCTZ) given to diabetic patients with stage 2 systolic hypertension (mean sitting systolic blood pressure (msSBP) ≥ 160 mm Hg and < 200 mm Hg).

ELIGIBILITY:
Inclusion criteria:

1. Male or female outpatients ≥ 18 years old.
2. Patients with a diagnosis of stage 2 hypertension (defined as an office cuff msSBP ≥ 160 mmHg and < 200 mmHg) at Visit 5 (randomization).
3. Patients with diabetes mellitus (Type 2) with an HbA1c at visit 1 ≤ 9.0 % and currently on stable anti-diabetic regimen or stable diet and exercise for at least 4 weeks prior to visit 1.
4. Patients who are eligible and able to participate in the study, and who are willing to give written informed consent before any assessment is performed.

Exclusion criteria:

1. Office blood pressure measured by cuff (msSBP ≥ 200 mmHg or msDBP ≥ 110 mmHg) at Visits 1-5.
2. History or evidence of secondary hypertension of any etiology (e.g., uncorrected renal artery stenosis, pheochromocytoma).
3. History of hypertensive encephalopathy or heart failure (NYHA Class II-IV).
4. Cerebrovascular accident, transient ischemic cerebral attack (TIA), coronary bypass surgery, myocardial infarction or any percutaneous coronary intervention (PCI) within 1 year prior to Visit 1.
5. Serum sodium less than the lower limit of normal, serum potassium < 3.5 mEq/L (corresponding to 3.5 mmol/L) or ≥ 5.3 mEq/L (corresponding to 5.3 mmol/L), or dehydration at Visit 1.
6. Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive hCG laboratory test (> 5 mIU/mL).
7. Use of other investigational drugs within 30 days of enrollment.
8. History of hypersensitivity to any of the study drugs or to drugs belonging to the same therapeutic class (thiazide diuretics, renin inhibitors, calcium channel blockers, or dihydropyridine like calcium channel blockers) as the study drugs.
9. History of gouty arthritis.
10. Long QT syndrome or QTc > 450 msec for males and > 470 msec for females at screening.
11. History of malignancy of any organ system (other than localized basal cell carcinoma of the skin), treated or untreated, within the past 5 years, regardless of whether there is evidence of local recurrence or metastases.
12. Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant including women whose career, lifestyle, or sexual orientation precludes intercourse with a male partner and women whose partners have been sterilized by vasectomy or other means, UNLESS they are using two birth control methods. The two methods can be a double barrier method or a barrier method plus a hormonal method.

    * Adequate barrier methods of contraception include: diaphragm, condom (by the partner), intrauterine device (copper or hormonal), sponge or spermicide. Hormonal contraceptives include any marketed contraceptive agent that includes an estrogen and/or a progestational agent. Reliable contraception should be maintained throughout the study and for 7 days after study drug discontinuation.
    * Women are considered post-menopausal and not of child bearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g. age appropriate, history of vasomotor symptoms) or six months of spontaneous amenorrhea with serum FSH levels > 40 mIU/mL (and estradiol< 20 pg/mL) or have had surgical bilateral oophorectomy (with or without hysterectomy) at least six weeks ago. In the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment.
13. Known Keith-Wagener grade III or IV hypertensive retinopathy.
14. Current angina pectoris requiring pharmacological therapy (except sublingual nitroglycerin).
15. Second or third degree heart block without a pacemaker.
16. Atrial fibrillation or atrial flutter at Visit 1, or potentially life-threatening or any symptomatic arrhythmia during the 12 months prior to Visit 1.
17. Clinically significant valvular heart disease.
18. History of angioedema during use of an ACE inhibitor.
19. History or evidence of drug or alcohol abuse within the last 12 months.
20. Any surgical or medical condition, which in the opinion of the investigator, may place the patient at higher risk from his/her participation in the study, or is likely to prevent the patient from complying with the requirements of the study or completing the study.
21. Any surgical or medical condition which might significantly alter the absorption, distribution, metabolism, or excretion of study drugs including, but not limited to, any of the following:

    * History of major gastrointestinal tract surgery such as gastrectomy, gastroenterostomy, or bowel resection.
    * History of active inflammatory bowel disease during the 12 months prior to Visit 1.
    * Currently active gastritis, duodenal or gastric ulcers, or gastrointestinal bleeding during the 3 months prior to Visit 1.
    * Any history of pancreatic injury, pancreatitis, or evidence of impaired pancreatic function/injury as indicated by abnormal lipase or amylase during the 12 months prior to Visit 1.
    * Evidence of hepatic disease as determined by any one of the following: ALT or AST values exceeding 3 x ULN at Visit 1, a history of hepatic encephalopathy, a history of esophageal varices, or a history of portocaval shunt.
    * Evidence of renal impairment as determined by any one of the following: serum creatinine > 1.5 x ULN at Visit 1, a history of dialysis, or a history of nephrotic syndrome.
    * Current treatment with cholestyramine or colestipol resins
22. History of noncompliance to medical regimes or unwillingness to comply with the study protocol.
23. Any condition that in the opinion of the investigator would confound the evaluation and interpretation of efficacy and/or safety data.
24. Persons directly involved in the execution of this protocol.
25. Known contraindications to the study drugs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 860 (Actual)
Dates: Start 2008-11; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Study Chair — Novartis
Locations (1):
- Sites in USA, East Hanover, New Jersey, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Aliskiren/HCTZ: Aliskiren / HCTZ 150/12.5 mg for 1 week followed by 300/25 mg for 7 weeks
- Amlodipine: Amlodipine 5 mg for 1 week followed by 10 mg for 7 weeks
Period: Overall Study
Arm/Group | Aliskiren/HCTZ | Amlodipine
Started | 428 | 432
Completed | 382 | 376
Not Completed | 46 | 56
Not completed — Administrative Problems | 3 | 0
Not completed — Adverse Event | 14 | 25
Not completed — Lost to Follow-up | 3 | 6
Not completed — Protocol Violation | 7 | 3
Not completed — Withdrawal by Subject | 6 | 13
Not completed — Lack of Efficacy | 13 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Aliskiren/HCTZ | Amlodipine | Total
Number analyzed (Participants) | 428 | 432 | 860
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.7 (9.83) | 59.8 (10.01) | 59.8 (9.91)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 212 | 209 | 421
  Male | 216 | 223 | 439

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Mean Sitting Systolic Blood Pressure (msSBP)
Time Frame: Baseline and Week 8
Population: Full analysis set, intent-to-treat
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Aliskiren/HCTZ | Amlodipine
Number analyzed (Participants) | 426 | 429
mmHg | -28.82 (0.722) | -26.22 (0.719)

2. Secondary Outcome: Change From Baseline in Mean Sitting Diastolic Blood Pressure (msDBP)
Time Frame: Baseline and Week 8
Population: Full analysis set, intent-to-treat
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Aliskiren/HCTZ | Amlodipine
Number analyzed (Participants) | 426 | 429
mmHg | -9.92 (0.414) | -8.97 (0.412)

3. Secondary Outcome: Percentage of Responders
Description: Response defined by mean sitting Systolic Blood Pressure < 130 mm Hg or a reduction of mean sitting Systolic Blood Pressure >= 20 mm Hg from baseline
Time Frame: Week 8
Population: Full analysis set, intent-to-treat
Measure: Number; unit: Percentage of Participants
Arm/Group | Aliskiren/HCTZ | Amlodipine
Number analyzed (Participants) | 426 | 429
Percentage of Participants | 74.2 | 68.5

4. Secondary Outcome: Percentage of Patients Achieving Blood Pressure Control
Description: Blood pressure control is defined as patient achieving a target Blood Pressure of mean sitting Systolic BloodPressure / mean sitting Diastolic Blood Pressure < 130/80 mmHg.
Time Frame: after 8 weeks of treatment
Population: Full analysis set, intent-to-treat
Measure: Number; unit: Percentage of Participants
Arm/Group | Aliskiren/HCTZ | Amlodipine
Number analyzed (Participants) | 426 | 429
Percentage of Participants | 23.2 | 13.8

5. Secondary Outcome: Biomarker Measurements
Description: Geometric mean of the post to baseline ratio in biomarkers of plasma renin activity (ng/ml/h), plasma renin concentration (ng/L), and cystatin C (mg/L)
Time Frame: Baseline and Week 8
Population: Full analysis set, intent-to-treat
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Aliskiren/HCTZ | Amlodipine
Number analyzed (Participants) | 428 | 432
ratio
  Plasma Renin activity (ng/ml/h) (N= 317, 300) | 0.42 (2.41) [0.37 to 0.48] | 1.75 (2.10) [1.57 to 1.94]
  Plasma Renin concentration (ng/L) (N=315, 299) | 9.53 (189.75) [8.32 to 10.91] | 1.49 (21.59) [1.36 to 1.62]
  Cystatin C (mg/L) (N = 327 , 310) | 1.04 (0.15) [1.03 to 1.06] | 0.98 (0.09) [0.97 to 0.99]

6. Secondary Outcome: Evaluate the Safety and Tolerability
Description: Percentage of patients with Adverse Event and percentage of patients with edema
Time Frame: after 8 weeks of treatment
Population: safety
Measure: Number; unit: Percentage of participants
Arm/Group | Aliskiren/HCTZ | Amlodipine
Number analyzed (Participants) | 428 | 431
Percentage of participants
  Any Adverse Event | 36.0 | 48.3
  edema | 2.6 | 17.6

ADVERSE EVENTS:
Arm/Group | Aliskiren/HCTZ | Amlodipine
Serious Adverse Events (participants affected / at risk) | 3/428 | 4/431
Other Adverse Events (participants affected / at risk) | 28/428 | 86/431
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Aliskiren/HCTZ (N=428) | Amlodipine (N=431)
Angina pectoris (Cardiac disorders) | 0 | 1
Angina unstable (Cardiac disorders) | 1 | 0
Coronary artery disease (Cardiac disorders) | 0 | 1
Myocardial ischaemia (Cardiac disorders) | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 2
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Aliskiren/HCTZ (N=428) | Amlodipine (N=431)
Oedema peripheral (General disorders) | 9 | 70
Headache (Nervous system disorders) | 19 | 22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial; or the publication of the trial results in their entirety.